CLINICAL TRIAL: NCT02996461
Title: VRC 320: A Phase I, Randomized Clinical Trial to Evaluate the Safety and Immunogenicity of a Zika Virus DNA Vaccine, VRC-ZKADNA090-00-VP, Administered Via Needle and Syringe or Needle-free Injector, PharmaJet, in Healthy Adults
Brief Title: VRC 320: A Phase I, Randomized Clinical Trial to Evaluate the Safety and Immunogenicity of a Zika Virus DNA Vaccine, VRC-ZKADNA090-00-VP, Administered Via Needle and Syringe or Needle-free Injector, PharmaJet, inHealthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 170024; 17-I-0024
Record Dates: First submitted 2016-12-16; First posted 2016-12-19 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-09-03

CONDITIONS: Prevention of Zika Infection; Zika-Specific Immune Response
Keywords: Zika Infection; Immune Response; Flavivirus; Arthropod-Borne Virus

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (3):
- Group 1 (Experimental): ZIKV DNA vaccine administered IM via needle and syringe at a single dosage of 4 mg on Day 0, week 4 and week 8.
  Interventions: Biological: VRC-ZKADNA090-00-VP
- Group 2 (Experimental): ZIKV DNA vaccine administered IM via needle and syringe as a split dose of two .5 ml injections on Day 0, week 4 and week 8.
  Interventions: Biological: VRC-ZKADNA090-00-VP
- Group 3 (Experimental): ZIKV DNA vaccine administered IM via needle-free injection device, PharmaJet, as a split dose of two .5 ml injections on Day 0, week 4 and week 8.
  Interventions: Biological: VRC-ZKADNA090-00-VP

INTERVENTIONS:
Biological: VRC-ZKADNA090-00-VP — VRC-ZKADNA090-00-VP is an investigational ZIKV DNA vaccine that is intended to prevent Zika virus infection.

SUMMARY:
Background:

People get Zika virus from infected mosquitos. They usually don t get very sick. But birth defects were reported in babies born to mothers who had Zika infection. In rare cases, people with Zika infection had a nervous system disease that causes severe muscle weakness and can be life threatening. A new vaccine made from DNA in the code for a Zika virus protein could help the body build an immune response against the virus.

Objectives:

To see if a new vaccine against Zika virus disease is safe and causes any side effects. To study specific immune responses to the vaccine.

Eligibility:

Healthy people ages 18-50

Design:

Participants will be screened with:

Medical history

Physical exam

Urine tests

Participants will have 18 visits over 2 years.

Participants will be randomly assigned to 1 of 3 groups. All will get 3 vaccines at 3 separate monthly visits. They will receive the vaccine in the upper arm muscle. Some will get it by needle and syringe, others by a device that uses high pressure to push the vaccine through the skin.

Vaccine visits last 4-6 hours. Participants will get a thermometer to measure their temperature and a ruler to measure any skin changes at the injection site. They will record this data for 7 days after each injection.

Other visits last 1-2 hours. These include:

Evaluation of any health changes or problems

Blood tests: Some samples may be used for future research.

Participants with side effects may have extra visits.

...

DETAILED DESCRIPTION:
STUDY DESIGN:

This is a Phase I, randomized clinical study to evaluate the safety, tolerability, and immunogenicity of a 3 dose vaccination regimen with the Zika virus (ZIKVwt) DNA vaccine, VRC-ZKADNA090-00-VP. Subjects will be randomized to one of three groups to receive a full 4 mg dose: 1) full dose by one intramuscular (IM) injection with needle and syringe; 2) split dose given as two 0.5 mL IM injections with needle and syringe; 3) split dose given as two 0.5 mL IM injections with PharmaJet, a needle-free injection device. The primary hypothesis is that the investigational ZIKVwt DNA vaccine will be safe and well tolerated in healthy adults. A secondary hypothesis is that the vaccine will elicit a ZIKV-specific immune response. The primary objectives are to evaluate the safety and tolerability of the vaccine in healthy adults. Secondary objectives are related to the immunogenicity of the vaccine and vaccination regimens.

PRODUCT DESCRIPTION:

The investigational vaccine, VRC-ZKADNA090-00-VP, was developed by the Vaccine Research Center (VRC), National Institute of Allergy and Infectious Diseases (NIAID), National Institutes of Health (NIH) and is composed of a single closed-circular DNA plasmid (VRC 5283) that encodes the wild type (wt) precursor membrane M (prM) and envelope (E) proteins from the H/PF/2013 strain of ZIKV. ZIKVwt

SUBJECTS:

Healthy adults 18 to 50 years of age.

STUDY PLAN:

Forty-five subjects will be enrolled at the NIH Clinical Center and randomized to 3 groups to receive study product on Day 0, Week 4 and Week 8. The protocol requires about 18 scheduled clinic visits and a telephone follow-up contact after each study product administration. Solicited reactogenicity will be evaluated using a 7-day diary card. Assessment of vaccine safety will include clinical observation and monitoring of hematological and chemical parameters at clinical visits throughout the study.

VRC 320 STUDY SCHEMA:

* Group 1:

  * Administration Method = Single Dose Needle and Syringe;
  * Subjects = 15;
  * Administration Schedule = Day 0 (ZIKVwt DNA(1 (1 mL) injection)), Week 4 (ZIKVwt DNA (1 (1 mL) injection)), Week 8 (ZIKVwt DNA (1 (1 mL) injection))
* Group 2:

  * Administration Method = Split Dose Needle and Syringe;
  * Subjects = 15;
  * Administration Schedule = Day 0 (ZIKVwt DNA(2 (0.5 mL) injections)), Week 4 (ZIKVwt DNA (2 (0.5 mL) injections)), Week 8 (ZIKVwt DNA (2 (0.5 mL) injections))
* Group 3:

  * Administration Method = Split Dose PharmaJet;
  * Subjects = 15;
  * Administration Schedule = Day 0 (ZIKVwt DNA(2 (0.5 mL) injections)), Week 4 (ZIKVwt DNA (2 (0.5 mL) injections)), Week 8 (ZIKVwt DNA (2 (0.5 mL) injections))
  * Subjects Total = 45 (All injections total a dose of 4 mg. ** Up to 50 total enrollments are permitted if additional subjects are needed to assess safety or immunogenicity.)

STUDY DURATION:

Subjects will be evaluated for safety and immune responses throughout the study for 44 weeks following the first vaccine administration. Durability of immune responses will be evaluated at two long term follow-up visits, occurring at 18 and 24 months

ELIGIBILITY:
* INCLUSION CRITERIA:

A subject must meet all of the following criteria:

* 18 to 50 years old
* Available for clinic visits for 24 months after enrollment
* Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
* Able and willing to complete the informed consent process
* Willing to donate blood for sample storage to be used for future research
* In good general health without clinically significant medical history
* Physical examination and laboratory results without clinically significant findings and a Body Mass Index (BMI) less than or equal to 40 within the 56 days prior to enrollment
* Agrees not to receive licensed or investigational flavivirus vaccines through 4 weeks after last product administration
* Laboratory Criteria within 56 days prior to enrollment:

  * Hemoglobin within institutional normal limits or accompanied by the site Principal Investigator (PI) or designee approval
  * WBC and differential either within institutional normal range or accompanied by site PI or designee approval
  * Total lymphocyte count greater than or equal to 800 cells/mm^3
  * Platelets = 125,000 - 500,000/mm^3
  * Alanine aminotransferase (ALT) less than or equal to 1.25 x institutional upper limit of normal (ULN)
  * Serum creatinine less than or equal to 1.1 x institutional ULN
  * Negative for HIV infection by an FDA approved method of detection
* Criteria applicable to women of childbearing potential:

  * Negative human chorionic gonadotropin (beta-HCG) pregnancy test (urine or serum) on day of enrollment
  * Agrees to use an effective means of birth control from at least 21 days prior to enrollment through 12 weeks after the last study vaccination

EXCLUSION CRITERIA:

A subject will be excluded if one or more of the following conditions apply:

* Female-specific: Breast-feeding or planning to become pregnant while participating through 12 weeks after the last study vaccination
* Subject has received any of the following:

  * More than 10 days of systemic immunosuppressive medications or cytotoxic medications within the 4 weeks prior to enrollment or any within the 14 days prior to enrollment
  * Blood products within 16 weeks prior to enrollment
  * Inactivated vaccines within 2 weeks prior to enrollment
  * Live attenuated vaccines within 4 weeks prior to enrollment
  * Investigational research products within 4 weeks prior to enrollment or planning to receive investigational products while on the study
  * Current allergen immunotherapy with antigen injections, unless on maintenance schedule
  * Current anti-TB prophylaxis or therapy
* Subject has a history of any of the following clinically significant conditions:

  * Laboratory confirmed ZIKV infection by self-report at the time of enrollment
  * Serious reactions to vaccines that preclude receipt of study vaccinations as determined by the site investigator
  * Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema
  * Asthma that is not well controlled
  * Diabetes mellitus (type I or II), with the exception of gestational diabetes
  * Evidence of autoimmune disease or immunodeficiency
  * Idiopathic urticaria within the past year
  * Hypertension that is not well controlled
  * Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
  * Malignancy that is active or history of malignancy that is likely to recur during the period of the study
  * Seizure disorder other than: 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures that have not required treatment within the last 3 years
  * Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen
  * Guillain-Barre Syndrome, Bell's palsy or similar neurological conditions
  * Psychiatric condition that precludes compliance with the protocol; past or present psychoses; or within 5 years prior to enrollment, a history of suicide plan or attempt
  * Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2016-12-12; Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of v ZIKV DNA vaccine administered at 4mg IM by needle and syringe. | Through 44 weeks of study participation.
To evaluate the safety and tolerability of ZIKV DNA vaccine administered at 4 mg IM by Pharma jet. | Through 44 weeks of study participation.

SECONDARY OUTCOMES:
To evaluate the magnitude and the frequency of ZIKV-specific antibody response as measured by neutralization assay. | Four weeks after the first, second and third injections for each regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Grace L Chen, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Dowd KA, Ko SY, Morabito KM, Yang ES, Pelc RS, DeMaso CR, Castilho LR, Abbink P, Boyd M, Nityanandam R, Gordon DN, Gallagher JR, Chen X, Todd JP, Tsybovsky Y, Harris A, Huang YS, Higgs S, Vanlandingham DL, Andersen H, Lewis MG, De La Barrera R, Eckels KH, Jarman RG, Nason MC, Barouch DH, Roederer M, Kong WP, Mascola JR, Pierson TC, Graham BS. Rapid development of a DNA vaccine for Zika virus. Science. 2016 Oct 14;354(6309):237-240. doi: 10.1126/science.aai9137. Epub 2016 Sep 22. PMID 27708058
- [Background] Ledgerwood JE, Graham BS. DNA vaccines: a safe and efficient platform technology for responding to emerging infectious diseases. Hum Vaccin. 2009 Sep;5(9):623-6. doi: 10.4161/hv.8627. No abstract available. PMID 19779298
- [Background] Graham BS, Ledgerwood JE, Nabel GJ. Vaccine development in the twenty-first century: changing paradigms for elusive viruses. Clin Pharmacol Ther. 2009 Sep;86(3):234-6. doi: 10.1038/clpt.2009.128. PMID 19707212
- [Derived] Gaudinski MR, Houser KV, Morabito KM, Hu Z, Yamshchikov G, Rothwell RS, Berkowitz N, Mendoza F, Saunders JG, Novik L, Hendel CS, Holman LA, Gordon IJ, Cox JH, Edupuganti S, McArthur MA, Rouphael NG, Lyke KE, Cummings GE, Sitar S, Bailer RT, Foreman BM, Burgomaster K, Pelc RS, Gordon DN, DeMaso CR, Dowd KA, Laurencot C, Schwartz RM, Mascola JR, Graham BS, Pierson TC, Ledgerwood JE, Chen GL; VRC 319; VRC 320 study teams. Safety, tolerability, and immunogenicity of two Zika virus DNA vaccine candidates in healthy adults: randomised, open-label, phase 1 clinical trials. Lancet. 2018 Feb 10;391(10120):552-562. doi: 10.1016/S0140-6736(17)33105-7. Epub 2017 Dec 5. PMID 29217376